## **Consent form template**

The consent form template below will be suitable for many studies but may need alterations to be commensurate with your study and must be used in conjunction with the guidance given in *Information Sheets & Consent Forms. Guidance for Researchers and Reviewers* 

For some studies a fuller, itemised or hierarchical consent form may be needed to cover important issues, especially if additional elements are optional for the participant. These may include:

- additional invasive tests or samples required for study purposes only;
- consent to use of audio/video-taping, with possible use of verbatim quotation or use of photographs;
- transfer of data/samples to countries with less data protection;
- agreement to receive individual feedback from testing.

| Centre Number: | | | |
|---|---|---|---|
| Stu | dy Number: IRAS Num. 196031 | | |
| Pat | ient Identification Number for this trial: | | |
| | CONSENT FORM FOR HEALTHY V | OLUNTEERS | _ |
| Titl | e of Project: | | |
| | Serum blood clotting changes during blood sampling v | ia non-luer one way filter valve | |
| | intravenous needle: Implications on the epidural | l blood patch procedure | |
| Na | me of Researcher: Dr Paul Sharpe | Please initial all boxe | s |
| 1. | I confirm that I have read and understand the information sh (version [2]) for the above study. I have had the opportunity ask questions and have had these answered satisfactorily. | | _ |
| 2. | I understand that my participation is voluntary and that I am free to withdraw at any time without giving any reason, without my medical care or legal rights being affected. | | |
| 3. | I agree for the research team to take blood samples from me with needles for the purposes of this study | | |
| 4. | . I agree to my GP being informed if any abnormalities are found . | | |
| 5. | I agree to take part in the above study. | | |
| | ne of Participant Date | Signature | |

Signature

Date

Name of person taking consent.